CLINICAL TRIAL: NCT01623219
Title: Community-Based Telemedicine to Reduce Risk to Georgia Veterans With PTSD
Brief Title: Community-Based Telemedicine to Reduce Risk to Georgia Veterans With Post Traumatic Stress Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Barbara O. Rothbaum, PhD, Professor in Psychiatry and Associate Vice Chair of Clinical Research, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00055554; Telemedicine_ECIC_2012 (Other: Other)
Record Dates: First submitted 2012-06-12; First posted 2012-06-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Post Traumatic Stress Disorder, PTSD
Keywords: PTSD; trauma; combat trauma; veterans; telemedicine; prolonged exposure
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TeleMedicine Prolonged Exposure (Experimental): Veterans will receive prolonged exposure therapy (PE)delivered via telemedicine instead of in person. For this study 9 weekly 90 minute sessions will be given over a period of up to 3 months. The first 2 sessions of each treatment will involve education, rational and treatment preparation. Sessions 3-9 will consist of recounting the traumatic event out loud and repeatedly. The purpose of this study is to determine if this treatment is effective when given through telehealth.
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — Exposure therapy refers to several cognitive behavioral treatment programs that involve confronting feared but safe thoughts, images, objects, situations, or activities in order to reduce unrealistic fear and anxiety. Exposure therapy for PTSD involves prolonged, imaginal exposure to the patient's traumatic memory and in vivo (in real life) exposure to trauma reminders. Prolonged exposure (PE) is a specific exposure therapy program that consists of five components: (1) psychoeducation (2) training in controlled breathing, (3) prolonged imaginal exposure to the trauma memory conducted in therapy sessions and repeated as homework, (4) prolonged in vivo exposure implemented as homework, and (5) processing of the traumatic material to correct maladaptive cognitions.
  Other Names: PE; Exposure Therapy; Imaginal Exposure

SUMMARY:
The investigator proposes to examine treatment for Posttraumatic Stress Disorder for Veterans who served in Iraq and Afghanistan provided through telemedicine which connects patients to doctors in different locations using the internet. In this study, Veterans will receive prolonged exposure therapy (PE). This treatment has been shown to be effective in reducing PTSD symptoms. For this study 9 weekly 90 minute sessions will be given over a period of up to 3 months. The first 2 sessions of each treatment will involve education, rational and treatment preparation. Sessions 3-9 will consist of recounting the traumatic event out loud and repeatedly. The purpose of this study is to determine if this treatment is effective when given through telehealth. To this end, the investigators propose to enroll up to 20 individuals who will access the investigators services through the GA telehealth network who has hundreds of telehealth sites across the state of Georgia. Patients will go to these sites to access the investigators therapists using GA telehealth equipment. The investigators hypothesize that PE delivered remotely through telemedicine will work to reduce the symptoms of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet DSM-IV criteria for PTSD due to exposure to a trauma while serving in Operation Iraqi Freedom, Operation Enduring Freedom-Afghanistan, and/or Operation New Dawn.
* Patients must be literate in English.
* Patients must be medically healthy or medically stable such that the stress of the therapy is not contraindicated.
* Participants must comprehend his or her role in treatment and the risks involved in order to be entered.

Exclusion Criteria:

* Patients with a history of mania, schizophrenia, or other psychoses
* Patients with prominent suicidal ideation
* Patients with current alcohol or drug dependence
* Patients with special medical conditions such as pregnancy, renal insufficiency, those with various chronic diseases or a history of significant head injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
CAPS-Clinician Administered PTSD Scale | Post-Treatment (10 weeks)

SECONDARY OUTCOMES:
BDI-II-Beck Depression Inventory-II | Post-Treatment (10 weeks)
Credibility/Expectancy Questionnaire-CEQ | post treatment (10 weeks)
Client Satisfaction Questionnaire-CSQ | post treatment (10 weeks)
PTSD Symptom Scale Self Report-PSS-SR | Post-Treatment (10 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O Rothbaum, PhD, ABPP, Principal Investigator — Emory University, School of Medicine, Dept. of Psychiatry